CLINICAL TRIAL: NCT02879201
Title: Continuous Venovenous Hemodiafiltration Versus Sustained Low-efficiency Hemodialysis for Critically Ill Patients With Acute Kidney Injury in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 036/59; Vajira002 (Registry Identifier: SLED)
Record Dates: First submitted 2016-07-25; First posted 2016-08-25 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Slow efficiency dialysis (Active Comparator): SLED is a kind of hemodialysis technique performed using Fresenius 4008B dialysis machine with FDX 120 GW (NIKKISO Japan) dialyzer. SLED sessions were 6-8 hour duration, three times per week (except Sunday), In case of severe volume overload, the session could be increased to meet clinical situation. Blood flow was maintained between 150-200 mL/hr and the dialysate flow of 300 mL/hr. Both the groups use unfractionated heparin as anticoagulant to prevent clotting of the extracorporeal circuit .the target partial thromboplastin time( PTT) was not more than twice the control level.
  Interventions: Procedure: Slow efficiency dialysis
- Continuous renal replacement therapy (No Intervention): CRRT is a kind of therapy involved continuos dialysis throughout 24 hours by using Edward Delivery system (Edward Life Science) as continuous venovenous hemodiafiltration (CVVHDF) mode using Aquamax HF 12 dialyzer. Blood flow rate was kept from 100-200 mL/hr and target effluent rates of 20 mL/hr . The substitution fluid was infused at a rate of 1,000 ml/hr with ultrafiltration rate at 100-300 mL/hr.Intervention here is the different mode of dialysis

INTERVENTIONS:
Procedure: Slow efficiency dialysis — Slow dialysis 4 times weekly 8 hours CVVHDF predilution mode
  Other Names: CRRT
  Arms: Slow efficiency dialysis

SUMMARY:
The investigators conducted a comparison trial between SLED and CRRT in critically ill patients to evaluate the outcome for all cause mortality at 30 day . The secondary outcome were recovery of renal function, complications during therapy and duration of hospitalization.

DETAILED DESCRIPTION:
The investigators performed a single center experience accumulated over 12 months since February 2009 with a continuous venovenous hemodiafiltration (CVVHDF) and hybrid technique named sustained low-efficiency dialysis (SLED). The primary end point was death from any cause by day 30. Intensive care unit (ICU) patients were eligible for inclusion when serum creatinine was > 2 mg/dL, and renal replacement therapy (RRT) was initiated. The selected patients were treated with CVVHDF or SLED.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria were

1. AKI requiring RRT
2. Hemodynamic instability defined by systolic blood pressure ≤ 90 mmHg and/or diastolic blood pressure ≤ 60 mmHg
3. Patients requiring initiation to vasopressor support

Exclusion Criteria:

* Patients with pre-existing chronic kidney disease ( eGFR less than 30 mLmin/1.73m2) were excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 day
  ll-cause mortality at 30 days following RRT initiation

SECONDARY OUTCOMES:
Numbers of patients with abnormal laboratory values | 30 days
  Renal function impairment
ICU stay | 30 days
  Total days in ICU

OTHER OUTCOMES:
Adverse events during treatment | 30 days
  Number of patients with catheter infection

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Unit, BMA Medical College and Vajira Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manns B, Doig CJ, Lee H, Dean S, Tonelli M, Johnson D, Donaldson C. Cost of acute renal failure requiring dialysis in the intensive care unit: clinical and resource implications of renal recovery. Crit Care Med. 2003 Feb;31(2):449-55. doi: 10.1097/01.CCM.0000045182.90302.B3. PMID 12576950